CLINICAL TRIAL: NCT04954092
Title: An Open Label Study With an Open Dose Selection Period to Assess the Safety, Tolerability and Immunogenicity of the Drug "Gam-COVID-Vac, a Combined Vector Vaccine for the Prevention of Coronavirus Infection Caused by the SARS-CoV-2 Virus", With the Participation of Adolescent Volunteers
Brief Title: Study of Gam-COVID-Vac in Adolescents
Acronym: OLSTAD
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Moscow Healthcare Department (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OLSTAD
Record Dates: First submitted 2021-07-05; First posted 2021-07-08 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Covid19; Vaccine Preventable Disease
Keywords: rAd vector based vaccine; Sputnik; rAd26; rAd5; adolescent
MeSH Terms: conditions — COVID-19; Vaccine-Preventable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 1/10 of full adult dose (Experimental)
  Interventions: Biological: Gam-COVID-vac M
- 1/5 of full adult dose (Experimental)
  Interventions: Biological: Gam-COVID-vac M
- Selected dose for second stage of the trial (Experimental)
  Interventions: Biological: Gam-COVID-vac M
- Placebo for second stage of the trial (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Gam-COVID-vac M — The vaccine consists of two components: component I and component II. Component I includes a recombinant adenoviral vector based on human adenovirus serotype 26 carrying the gene for the S-protein of the SARS-CoV-2 virus, component II includes a vector based on human adenovirus serotype 5 carrying the protein S gene of the SARS-CoV-2 virus
  Arms: 1/10 of full adult dose; 1/5 of full adult dose; Selected dose for second stage of the trial
Biological: Placebo — Composition without active ingredients
  Arms: Placebo for second stage of the trial

SUMMARY:
Double-blind, placebo-controlled study with open dose selection period for safety assessment, tolerance and immunogenicity of the drug "GamKOVID-Vac M, a combined vector vaccine for prevention of coronavirus infection caused by the virus SARS-CoV-2" in adolescents

DETAILED DESCRIPTION:
The study will include healthy volunteers aged 12-17 years inclusive. Volunteers will be recruited in at least two clinical centers. Teams will be divided into subgroups to ensure the safety of volunteers during hospitalization amid the ongoing pandemic.

Stage 1 (Phase I-II) - 100 volunteers will be included in two dosing groups (50 in each group), a sufficient number of volunteers should be screened (no more than 7 days before inclusion in the study). To ensure the required number of volunteers who have completed screening procedures (pre-screening procedures can be organized).

The conditions of the study were the selection of doses (administration of the drug and observation for 48 hours) in a hospital setting, the rest of the visits were outpatient.

It is planned to start the study with a dose of 1/10 of the full adult dose. Volunteers will be hospitalized the day before vaccination. It is allowed to carry out screening procedures the day before vaccination in a hospital setting, subject to the prior approval of the volunteer based on the results of pre-screening. The first dose will be administered on day 1. After that, the volunteer will be monitored in the hospital for 48 hours. on days 3 and 7, a telephone consultation will be held. With a favorable safety profile after 7 days after the 1/10 dose, the Principal Investigators present a consolidated decision to escalate the dose to 1/5 of the adult dose on ICMD.

The transition to the next stage is planned on the basis of the report on the safety and tolerability of ILS on the 28th day after the introduction of the first component. The selected dose will be determined based on the immunogenicity scores at day 28, which should be consistent with the immunogenicity in adults after receiving the full dose of ILP.

Stage 2 (Phase III) - 3000 volunteers to be randomized to two groups - active drug and placebo in a ratio of 4: 1. Volunteers will receive the drug at the dose selected in the first phase. Research is carried out on an outpatient basis.

The randomization of research subjects will be carried out in two age strata: 12-14 years old and 15-17 years old.

The intramuscular vaccine will be administered at vaccination visits # 2 and # 3 (Day 1 and Day 21 ± 2) on an outpatient basis. After vaccination, TMK will be carried out for 2 days.

Follow-up visits # 4 (28 ± 2), 5 (42 ± 4), 6 (90 ± 7) and 7 (180 ± 14); TMK for 270 ± 14 and 365 ± 14 days.

Additionally historical control data will be used (data from phase III clinical trials of efficacy, safety and immunogenicity obtained during their evaluation in a sample of adult volunteers aged 18-21 years);

The duration of study participation for one subject will be 365 ± 14 days after the first dose of vaccine, during which each subject will undergo a screening visit, two hospitalizations for drug administration, five face-to-face visits to the investigator, and telephone contacts with the investigator.

The data of research subjects will be collected using electronic forms of individual registration cards, as well as using electronic questionnaires (diaries) filled in by research subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of written informed consent of the research subject and parents / adoptive parents of the subject to participate in the research;
2. Boys and girls aged 12-17 inclusive;
3. Negative test result for HIV, hepatitis, syphilis;
4. A negative test result for the presence of IgM and IgG antibodies to SARS CoV2 by enzyme immunoassay, as well as, if available, the result of an examination performed in medical institutions of the Moscow City Health Department 7 days prior to inclusion in the study can be taken into account;
5. A negative test result for COVID-2019, determined by the PCR method at the screening visit, and, if available, can be taken into account the result of the examination performed in the medical organizations of the Moscow City Health Department 7 days before being included in the study;
6. No history of COVID-2019;
7. Absence of contact of the research subject with COVID-2019 patients for at least 14 days prior to inclusion in the research (according to the research participant, parents / adoptive parents of the subject);
8. Consent to the use of effective contraceptive methods during the entire period of participation in the study;
9. Negative pregnancy test based on urine test results at the screening visit (for all girls - study participants);
10. Negative test for the presence of drugs and psychostimulants in the urine at the screening visit;
11. Negative alcohol test at screening visit;
12. No history of pronounced post-vaccination reactions or post-vaccination complications after the use of immunobiological drugs;
13. Absence of acute infectious and / or respiratory diseases for at least 14 days prior to enrollment in the study

Exclusion Criteria:

1. Any vaccination / immunization carried out within 30 days prior to enrollment in the study.
2. Therapy with steroids (with the exception of hormonal contraceptive drugs) and / or immunoglobulins or other blood products, not completed 30 days before enrollment in the study;
3. Immunosuppressive therapy and systemic therapy with corticosteroid drugs, completed in less than 3 months. prior to inclusion in the study.
4. Postponed acute coronary syndrome or stroke less than one year before inclusion in the study
5. Any immunodeficiency (for example, hereditary immunodeficiency, acquired immunodeficiency syndrome [AIDS], etc.).
6. Infectious diseases:

   * history of HIV (antibodies to HIV type 1 or 2), positive test for HBsAg or HCV RNA [qualitative]), active form of syphilis;
   * Tuberculosis;
   * Active infection (with the exception of onychomycosis), or any significant episode of infection requiring intravenous antibiotic treatment for 4 weeks before screening or by mouth for 2 weeks before screening;
   * A history of a serious recurrent or chronic infection not listed above.
7. Major surgery within 4 weeks prior to screening.
8. Chronic autoimmune diseases or systemic collagenoses in history, requiring the appointment of immunosuppressive therapy.
9. Volunteers who have undergone organ transplants, including bone marrow or peripheral blood stem cell (PBC) transplants, and are receiving immunosuppressive therapy.
10. History of splenectomy.
11. Volunteers with a previous or concomitant history of neoplasms (ICD codes C00-D09).
12. A burdened allergic history (history of anaphylactic shock, Quincke's edema and other life-threatening conditions), hypersensitivity or allergic reactions to the administration of immunobiological preparations, known allergic reactions to any component of a vaccine or vaccine containing similar components, exacerbation of allergic diseases on the day of inclusion in the study.
13. Neutropenia (decrease in the absolute number of neutrophils less than 1000 cells / mm3), agranulocytosis, significant blood loss, severe anemia (hemoglobin concentration less than 80 g / l), thrombocytopenia (decrease in the absolute number of platelets less than 50,000 cells / mm3).
14. Anorexia, protein deficiency of any origin.
15. Volunteers with a BMI <18 (low body weight) or a BMI ≥ 35 kg / m2.
16. Extensive tattoos at the injection sites (deltoid muscle area), which do not allow assessing the local response to the injection of ILP.
17. Chronic diseases of the cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of the gastrointestinal tract, liver, kidneys, muscle and connective tissue in the stage of exacerbation or decompensation.
18. Presence or suspicion of drug, alcohol or drug addiction and other mental disorders.
19. Diseases, the presence of which, from the point of view of the medical researcher, puts the health of the participant at risk if participating in the study or potentially complicates the interpretation of the results of the examination.
20. Family members of staff of research centers directly involved in the conduct of research, etc.
21. Participation in other clinical trials and use of other investigational drugs within 28 days of screening.
22. Planned vaccination against COVID-19 with any vaccine, both in the framework of other studies and in the framework of civil appeal.
23. Female subjects during pregnancy or lactation
24. Inability to read in Russian; inability or unwillingness to understand the essence of the research. Any other conditions that limit the eligibility of obtaining informed consent or that may affect the volunteer's ability to participate in the study affect the volunteer's ability to take part in the study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3000 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-11-06 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Geometric mean titer of antigen-specific IgGs | 21, 28, 42, 90, 180 days
  To define geometric mean titer of antigen-specific IgGs after vaccination
Geometric mean titer of neutralizing antibodies | 21, 28, 42, 90, 180 days
  To define geometric mean titer of neutralizing antibodies against SARS-Cov-2 virus after vaccination
IFN-gamma secretion by T lymphocytes | 21, 28, 42, 90, 180 days
  To define changes in level of IFN-gamma secretion by T lymphocytes under antigen stimulation
Frequency of adverse reactions | 365+/-14 days
  Frequency of vaccine-related adverse reactions
Severity of adverse reactions | 365+/-14 days
  Severity of vaccine-related adverse reactions

SECONDARY OUTCOMES:
Incidence of COVID-19 cases | within 28 to 365 days
  Incidence of mild, moderate, severe, extremely severe cases and deaths due to COVID-19

OTHER OUTCOMES:
Presence of anti-vector antibodies | before intervention and on 42, 180 days
  Presence of anti-rAd26 and anti-rAd5 antibodies before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Anna Vlasova, Principal Investigator — Morozovskaya Children's City Clinical Hospital of the Moscow Department of Health; Svetlana Borzakova, Principal Investigator — Children's City Clinical Hospital named after Z.A. Bashlyaeva of the Moscow Department of Health
Locations (2):
- Russia (2):
  - Children's City Clinical Hospital named after Z.A. Bashlyaeva of the Moscow Department of Health, Moscow
  - Morozovskaya Children's City Clinical Hospital of the Moscow Department of Health, Moscow

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tukhvatulin AI, Dolzhikova IV, Dzharullaeva AS, Grousova DM, Kovyrshina AV, Zubkova OV, Zorkov ID, Iliukhina AA, Shelkov AY, Erokhova AS, Popova O, Ozharovskaia TA, Zrelkin DI, Izhaeva FM, Shcheblyakov DV, Esmagambetov IB, Tokarskaya EA, Nikitenko NA, Lubenets NL, Khadorich EA, Gushchin VA, Borzakova SN, Vlasova AV, Osmanov IM, Gorev VV, Naroditsky BS, Logunov DY, Gintsburg AL. Safety and immunogenicity of rAd26 and rAd5 vector-based heterologous prime-boost COVID-19 vaccine against SARS-CoV-2 in healthy adolescents: an open-label, non-randomized, multicenter, phase 1/2, dose-escalation study. Front Immunol. 2023 Aug 1;14:1228461. doi: 10.3389/fimmu.2023.1228461. eCollection 2023. PMID 37600800